CLINICAL TRIAL: NCT03857035
Title: A PROSPECTIVE SPLIT MOUTH CLINICAL STUDY: OF PIEZOSURGERY AND CONVENTIONAL ROTARY INSTRUMENTS IN IMPACTED THIRD MOLAR SURGERY
Brief Title: COMPARISON OF PIEZOSURGERY AND CONVENTIONAL ROTARY INSTRUMENTS IN IMPACTED THIRD MOLAR SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Dilek Menziletoglu, Principle Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: NEU3
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-02

CONDITIONS: Impacted Third Molar Tooth
Keywords: Trismus; piezosurgery; pain; swelling
MeSH Terms: conditions — Trismus; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery group (Experimental): One side of the patients will be randomly selected and labeled as "experimental group". In experimental group, impacted third molar will be extracted using piezosurgery.
  Interventions: Other: Piezosurgery group
- Rotary Instruments Group (Placebo Comparator): The other side will be accepted as "control group". In the control group, impacted third molar will be extracted using conventional rotary instruments.
  Interventions: Other: Piezosurgery group

INTERVENTIONS:
Other: Piezosurgery group — Piezosurgery technique will be examined about impacted third molar surgery.

SUMMARY:
The purpose is to compare the effects of piezosurgery and conventional rotary instruments on postoperative pain, swelling, trismus and patients' comfort after mandibular third molar surgery.

DETAILED DESCRIPTION:
The investigators plan a prospective and split mouth study. Thirty patients will be randomly selected. Inclusion criteria were being older than 18 of age, having asymptomatic bilateral mesioangular impacted mandibular third molar (Pell and Gregory class II, position B) fully covered with mucosa and bone, and being otherwise medically healthy.

One side of the patients will be randomly selected and labeled as "experimental group". In experimental group, impacted third molar will be extracted using piezosurgery. The other side will be accepted as "control group". In the control group, impacted third molar will be extracted using conventional rotary instruments.There will at least one month between two surgeries. The investigators will compare postoperative pain, swelling, trismus and patients' comfort.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being older than 18 of age, having asymptomatic bilateral mesioangular impacted mandibular third molar (Pell and Gregory class II, position B) fully covered with mucosa and bone, and being otherwise medically healthy.

Exclusion Criteria:

* Exclusion criteria were as follows: Alcohol abuse, smoking, pregnancy, and presence of acute severe periodontitis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
All the patients will be given a form containing verbal rating scale ranging from 0 to 5, showing the degree of swelling. | Up to 1 week
  The edema measurement will be done during the one week after surgery.

SECONDARY OUTCOMES:
Pain will be assessed using a visual analogue scale. | Up to 1 week
  The level of postoperative pain will be evaluated using a 10-cm visual analogue scale , with zero representing no pain and 10 representing excruciating pain. Pain measurement will be done preoperatively, postoperative 2nd day, 7th day after the surgery.
Trismus will be evaluated using a caliper at maximum mouth opening. | Up to 1 week
  Trismus will be assessed by measuring the maximum interincisal opening (in millimetres) - the distance between the incisal margin of the upper and lower central incisors. Trismus measurement will be done preoperatively, postoperative 2nd day, 7th day after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, Dr, Principal Investigator — Necmettin Erbakan University
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Faculty of Dentistry, Konya, Karatay
  - Necmettin Erbakan University, Konya, Karatay

IPD SHARING:
Plan to Share IPD: No